CLINICAL TRIAL: NCT05714527
Title: Closed-Loop O2 Use During Invasive Mechanical Ventilation Of Pediatric Patients (CLOUDIMPP)- a Randomized Cross-over Study
Brief Title: Closed-Loop O2 Use During Invasive Mechanical Ventilation Of Pediatric Patients
Acronym: CLOUDIMPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Hasan ağın, Professor, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/750
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Failure
Keywords: Acute respiratory failure (ARF); Pediatric acute respiratory distress syndrome (PARDS); Closed-loop; Oxygen; SpO2
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close-loop FiO2 Controller (Experimental): Two hours period where the fraction of inspired oxygen (FiO2) delivered will be automatically titrated based on SpO2 values obtained from the patient.
  Interventions: Device: Close-loop FiO2 controller
- Conventional (Active Comparator): Conventional FiO2 adjustment by the clinician according to SpO2 values
  Interventions: Device: Conventional

INTERVENTIONS:
Device: Close-loop FiO2 controller — Close-loop FiO2 controller software option provides automated adjustment of the ventilator Oxygen setting to maintain the patient's SpO2 in a defined target range. When using the software option, the user defines the SpO2 target range, as well as the SpO2 emergency limits, and the device adjusts the FiO2 setting to keep the patient's SpO2 in the target range.
  Arms: Close-loop FiO2 Controller
Device: Conventional — Conventional FiO2 adjustment by the clinician according to SpO2 values, by using the manual FiO2 knob.
  Arms: Conventional

SUMMARY:
During mechanical ventilation (MV) hypoxemic or hyperoxemic events should be carefully monitored and a quick response should be provided by the caregiver at the bedside. Pediatric mechanical ventilation consensus conference (PEMVECC) guidelines suggest to measure SpO2 in all ventilated children and furthermore to measure partial arterial oxygen pressure (PaO2) in moderate-to-severe disease. There were no predefined upper and lower limits for oxygenation in pediatric guidelines, however, Pediatric acute lung injury consensus conference PALICC guidelines proposed SpO2 between 92 - 97% when positive end-expiratory pressure (PEEP) is smaller than 10 cm H2O and SpO2 of 88 - 92% when PEEP is bigger or equal to 10 cm H2O. For healthy lung, PEMVECC proposed the SpO2>95% when breathing a FiO2 of 21%. As a rule of thumb, the minimum fraction of inspired O2 (FiO2) to reach these targets should be used. A recent Meta-analyze showed that automated FiO2 adjustment provides a significant improvement of time in target saturations, reduces periods of hyperoxia, and severe hypoxia in preterm infants on positive pressure respiratory support. This study aims to compare the closed-loop FiO2 controller with conventional control of FiO2 during mechanical ventilation of pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients older than 1 month and younger than18 years of age; hospitalized at the PICU with the intention of treatment with IMV at least for the upcoming 5 hours
* Requiring FiO2 ≥ 25% to keep SpO2 in the target ranges defined by the clinician
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation

Exclusion Criteria:

* Patient with indication for immediate noninvasive ventilation (NIMV), High flow oxygen therapy (HFOT)
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Low quality on the SpO2 measurement using finger and ear sensor (quality index below 60% on the SpO2 sensor, which is displayed by a red or orange colour bar)
* Severe acidosis (pH ≤ 7.25)
* Pregnant woman
* Patients deemed at high risk for the need of non-invasive mechanical ventilation within the next 5 hours
* Patients deemed at high risk for the need of transportation from PICU to another ward, diagnostic unit or any other hospital
* Diseases or conditions which may affect transcutaneous SpO2 measurement such as chronic or acute dyshemoglobinemia: methemoglobinemia, carbon monoxide (CO) poisoning, sickle cell disease
* Formalized ethical decision to withhold or withdraw life support
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of acute respiratory failure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in optimal SpO2 range | 2 hours
  The optimal SpO2 range will be defined according to the SpO2 targets determined by the clinician.

SECONDARY OUTCOMES:
Percentage of time spent in suboptimal SpO2 range | 2 hours
  SpO2 values outside the optimal range but still within an acceptable limit (2-3 percent above and below the optimal range)
Mean FiO2 | 2 hours
  Mean fraction of inspired oxygen
Mean SpO2/FiO2 | 2 hours
  Mean SpO2/FiO2
Number of manual adjustments | 2 hours
  Frequency of manual adjustments of FiO2
Number of alarms | 2 hours
  Frequency of alarms
Percentage of time with SpO2 signal available | 2 hours
  Time with SpO2 signal available
Percentage of time with SpO2 below 88 and 85 percent | 2 hours
  Duration of time with SpO2 <85 percent and <88 percent, respectively
Number of events with SpO2 below 88 and 85 percent | 2 hours
  Frequency of SpO2 decreases <85 percent and <88 percent, respectively
Percentage of time with FiO2 below 40 percent, 60 percent and 100 percent | 2 hours
  Percentage of time that FiO2 is <40 percent, 60 percent and 100 percent, respectively
Total oxygen use | 2 hours
  Volume of total oxygen used (in L)

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Erzurum Regional Research and Training Hospital, Erzurum
  - Cam Sakura Research and Training Hospital, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kneyber MCJ, de Luca D, Calderini E, Jarreau PH, Javouhey E, Lopez-Herce J, Hammer J, Macrae D, Markhorst DG, Medina A, Pons-Odena M, Racca F, Wolf G, Biban P, Brierley J, Rimensberger PC; section Respiratory Failure of the European Society for Paediatric and Neonatal Intensive Care. Recommendations for mechanical ventilation of critically ill children from the Paediatric Mechanical Ventilation Consensus Conference (PEMVECC). Intensive Care Med. 2017 Dec;43(12):1764-1780. doi: 10.1007/s00134-017-4920-z. Epub 2017 Sep 22. PMID 28936698
- [Background] van Kaam AH, Hummler HD, Wilinska M, Swietlinski J, Lal MK, te Pas AB, Lista G, Gupta S, Fajardo CA, Onland W, Waitz M, Warakomska M, Cavigioli F, Bancalari E, Claure N, Bachman TE. Automated versus Manual Oxygen Control with Different Saturation Targets and Modes of Respiratory Support in Preterm Infants. J Pediatr. 2015 Sep;167(3):545-50.e1-2. doi: 10.1016/j.jpeds.2015.06.012. Epub 2015 Jul 2. PMID 26144575
- [Background] Lui K, Jones LJ, Foster JP, Davis PG, Ching SK, Oei JL, Osborn DA. Lower versus higher oxygen concentrations titrated to target oxygen saturations during resuscitation of preterm infants at birth. Cochrane Database Syst Rev. 2018 May 4;5(5):CD010239. doi: 10.1002/14651858.CD010239.pub2. PMID 29726010
- [Background] Maiwald CA, Niemarkt HJ, Poets CF, Urschitz MS, Konig J, Hummler H, Bassler D, Engel C, Franz AR; FiO2-C Study Group. Effects of closed-loop automatic control of the inspiratory fraction of oxygen (FiO2-C) on outcome of extremely preterm infants - study protocol of a randomized controlled parallel group multicenter trial for safety and efficacy. BMC Pediatr. 2019 Oct 21;19(1):363. doi: 10.1186/s12887-019-1735-9. PMID 31630690
- [Background] Sandal O, Ceylan G, Topal S, Hepduman P, Colak M, Novotni D, Soydan E, Karaarslan U, Atakul G, Schultz MJ, Agin H. Closed-loop oxygen control improves oxygenation in pediatric patients under high-flow nasal oxygen-A randomized crossover study. Front Med (Lausanne). 2022 Nov 16;9:1046902. doi: 10.3389/fmed.2022.1046902. eCollection 2022. PMID 36465920
- [Derived] Atakul G, Ceylan G, Sandal O, Soydan E, Hepduman P, Colak M, Zimmermann JM, Novotni D, Karaarslan U, Topal S, Agin H. Closed-loop oxygen usage during invasive mechanical ventilation of pediatric patients (CLOUDIMPP): a randomized controlled cross-over study. Front Med (Lausanne). 2024 Sep 10;11:1426969. doi: 10.3389/fmed.2024.1426969. eCollection 2024. PMID 39318593